CLINICAL TRIAL: NCT02889133
Title: A Randomized Trial to Determine if RBCs From Donors With Iron Deficient Erythropoiesis Have Decreased Post-transfusion RBC Recovery and Whether Iron Repletion Improves Recovery
Brief Title: Donor Iron Deficiency Study - Red Blood Cells From Iron-deficient Donors: Recovery and Storage Quality
Acronym: DIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: New York Blood Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eldad Arie Hod, Associate Professor of Pathology and Cell Biology, Dept of Pathology&Cell Biology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AAAQ8875; 1R01HL133049-01 (NIH)
Record Dates: First submitted 2016-08-25; First posted 2016-09-05 (Estimated); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Iron Deficiency
Keywords: Iron deficiency; Transfusion; Blood donation
MeSH Terms: conditions — Iron Deficiencies | interventions — Iron-Dextran Complex; Sodium Chloride; Saline Solution; Blood Donation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron repletion (Active Comparator): Subjects will donate blood donation and undergo 24-hour PTR and receive IV iron-dextran. After 5 months, subjects will donate blood again, receive IV saline and undergo 24-hour PTR.
  Interventions: Drug: Iron-dextran; Drug: Saline; Procedure: Blood Donation; Procedure: 24-hour PTR
- Placebo (Placebo Comparator): Subjects will donate blood donation and undergo 24-hour PTR and receive IV saline. After 5 months, subjects will donate blood again, receive IV iron-dextran and undergo 24-hour PTR.
  Interventions: Drug: Iron-dextran; Drug: Saline; Procedure: Blood Donation; Procedure: 24-hour PTR

INTERVENTIONS:
Drug: Iron-dextran — Approved for clinical use: 1-gram dose IV - diluted in 500 mL, one pint normal saline.
  Other Names: INFeD; Low molecular weight iron-dextran
Drug: Saline — Salt water IV - 500 mL, one pint normal saline.
  Other Names: Placebo; Normal Saline
Procedure: Blood Donation — Standard process of collecting and storing blood and blood components (approximately 450 mL, or a pint of blood). Following donation, the blood will be leukoreduced, packed, and stored in AS-3 solution.
  Other Names: Red blood cell donation
Procedure: 24-hour PTR — The way the FDA determines how good blood is for transfusion is called a "radioactive 51-Chromium 24-hour post-transfusion red cell recovery study." The purpose is to measure how many of the transfused red cells are still in circulation (being pumped by the heart through blood vessels) 24 hours after transfusion. In order to measure the percent of red cells that are still in circulation, a small amount of the donated blood will be radioactively labeled. This will be infused in one arm and then blood will be collected from the other arm at different time points to measure how much of the transfused red cells are still in circulation.
  Other Names: 24-hour post-transfusion red cell recovery

SUMMARY:
Primary Hypothesis

* The 24-hour post-transfusion RBC recovery of units obtained from donors exhibiting iron-deficient erythropoiesis will not meet FDA standards for clinical use.
* The 24-hour post-transfusion RBC recovery of units obtained after intravenous iron repletion will improve significantly and will meet FDA standards for clinical use.

DETAILED DESCRIPTION:
Iron deficiency is common among regular blood donors, but the recovery and quality of red blood cell (RBC) units from iron-deficient donors has not been rigorously examined. Evidence from both animal and human studies indicate that when the iron supply for erythropoiesis is inadequate, the RBCs produced have multiple metabolic defects that impair their ability to tolerate refrigerated storage. Studies in a mouse model demonstrated decreased post-transfusion recovery of refrigerator-stored RBCs obtained from iron-deficient donors. The planned studies will identify human donors at greatest risk of providing RBCs with poor post-transfusion recovery by using a combination of a decreased serum ferritin concentration and increased RBC zinc protoporphyrin, as described below. To evaluate unequivocally the role of iron deficiency in poor posttransfusion RBC recovery, intravenous iron will be used for iron repletion.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. healthy (by self report);
3. body weight >110 lbs;
4. female hematocrit >=38%, male hematocrit >39%;
5. frequent blood donor (men ≥2 and female ≥1 RBC unit donations in past year);
6. ferritin <=15 ng/mL; and
7. zinc protoporphyrin >=60 µmol/mol heme.

Exclusion Criteria:

1. ineligible for donation based on the New York Blood Center donor autologous questionnaire;
2. taking iron supplementation;
3. C-reactive protein >10 mg/L;
4. sickle cell trait;
5. systolic blood pressure >180 or <90 mm Hg, diastolic blood pressure >100 or <50 mm Hg;
6. heart rate <50 or >100;
7. temperature >99.5°F prior to donation;
8. temperature >100.4°F or subjective feeling of illness prior to 51-Chromium 24-hour RBC recovery study (to avoid the subject having a concurrent illness that may affect post-transfusion recovery);
9. positive results on standard blood donor infectious disease testing;
10. pregnancy;
11. taking, or planning to take, iron supplements; and
12. history of severe asthma requiring hospitalization, allergic eczema (atopic dermatitis), or other atopic allergy causing anaphylaxis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eldad A. Hod, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moroff G, Sohmer PR, Button LN. Proposed standardization of methods for determining the 24-hour survival of stored red cells. Transfusion. 1984 Mar-Apr;24(2):109-14. doi: 10.1046/j.1537-2995.1984.24284173339.x. PMID 6710582
- [Derived] Hod EA, Brittenham GM, Bitan ZC, Feit Y, Gaelen JI, La Carpia F, Sandoval LA, Zhou AT, Soffing M, Mintz A, Schwartz J, Eng C, Scotto M, Caccappolo E, Habeck C, Stern Y, McMahon DJ, Kessler DA, Shaz BH, Francis RO, Spitalnik SL. A randomized trial of blood donor iron repletion on red cell quality for transfusion and donor cognition and well-being. Blood. 2022 Dec 22;140(25):2730-2739. doi: 10.1182/blood.2022017288. PMID 36069596
- [Derived] Roussel C, Morel A, Dussiot M, Marin M, Colard M, Fricot-Monsinjon A, Martinez A, Chambrion C, Henry B, Casimir M, Volle G, Depond M, Dokmak S, Paye F, Sauvanet A, Le Van Kim C, Colin Y, Georgeault S, Roingeard P, Spitalnik SL, Ndour PA, Hermine O, Hod EA, Buffet PA, Amireault P. Rapid clearance of storage-induced microerythrocytes alters transfusion recovery. Blood. 2021 Apr 29;137(17):2285-2298. doi: 10.1182/blood.2020008563. PMID 33657208

RESULTS

PARTICIPANT FLOW:
Groups:
- Iron Repletion: Subjects will donate blood donation and undergo 24-hour PTR and receive IV iron-dextran. After 5 months, subjects will donate blood again and undergo 24-hour PTR.
  Iron-dextran: Approved for clinical use: 1-gram dose IV - diluted in 500 mL, one pint normal saline.
  Saline: Salt water IV - 500 mL, one pint normal saline.
  Blood Donation: Standard process of collecting and storing blood and blood components (approximately 450 mL, or a pint of blood). Following donation, the blood will be leukoreduced, packed, and stored in AS-3 solution.
  24-hour PTR: The way the FDA determines how good blood is for transfusion is called a "radioactive 51-Chromium 24-hour post-transfusion red cell recovery study." The purpose is to measure how many of the transfused red cells are still in circulation (being pumped by the heart through blood vessels) 24 hours after transfusion. In order to measure the percent of red cells that are still in circulation, a small amount of the donated blood will be radioactively labeled. This will be infused in one arm and then blood will be collected from the other arm at different time points to measure how much of the transfused red cells are still in circulation.
- Placebo: Subjects will donate blood donation and undergo 24-hour PTR and receive IV saline. After 5 months, subjects will donate blood again and undergo 24-hour PTR.
  Iron-dextran: Approved for clinical use: 1-gram dose IV - diluted in 500 mL, one pint normal saline.
  Saline: Salt water IV - 500 mL, one pint normal saline.
  Blood Donation: Standard process of collecting and storing blood and blood components (approximately 450 mL, or a pint of blood). Following donation, the blood will be leukoreduced, packed, and stored in AS-3 solution.
  24-hour PTR: The way the FDA determines how good blood is for transfusion is called a "radioactive 51-Chromium 24-hour post-transfusion red cell recovery study." The purpose is to measure how many of the transfused red cells are still in circulation (being pumped by the heart through blood vessels) 24 hours after transfusion. In order to measure the percent of red cells that are still in circulation, a small amount of the donated blood will be radioactively labeled. This will be infused in one arm and then blood will be collected from the other arm at different time points to measure how much of the transfused red cells are still in circulation.
Period: Completed Primary Outcome
Arm/Group | Iron Repletion | Placebo
Started | 39 | 40
Completed | 29 | 28
Not Completed | 10 | 12
Not completed — Lost to Follow-up | 1 | 1
Not completed — Manufacturing error | 3 | 8
Not completed — Chromium labeling failure | 1 | 0
Not completed — COVID-19/Illness | 4 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Subject did not meet donor criteria | 0 | 1
Period: Completed Secondary Outcomes
Arm/Group | Iron Repletion | Placebo
Started | 39 | 40
Completed | 33 | 35
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — COVID-19/illness | 4 | 2
Not completed — Subject could not donate blood after randomization | 0 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Repletion | Placebo | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [26 to 47] | 34 [26 to 49] | 34 [26 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 33 | 37 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 25 | 31 | 56
  More than one race | 7 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79
Weight [Median (Inter-Quartile Range); unit: kg] | 73 [64 to 79] | 66 [59 to 82] | 68 [60 to 82]

OUTCOME MEASURES:

1. Primary Outcome: 51-Chromium 24-hour Post-transfusion RBC Recovery of Units
Description: Comparison of the percentage change in 51-Chromium-labeled RBCs remaining from pre- and 24 hour post-transfusion measurement between the Iron Repletion and the Placebo group. The post-transfusion recovery represents the percent of 51-Chromium-labeled RBCs remaining in circulation 24 hours after infusion as compared to an extrapolated time zero measurement.
Time Frame: Performed 42 days after blood donation
Population: See participant flow for primary outcome for subject number explanation.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 29 | 28
percentage change | 1.6 [-0.5 to 3.8] | -0.4 [-2.0 to 1.2]

2. Secondary Outcome: RBC Zinc Protoporphyrin Levels
Description: Measured in a clinical laboratory. Will be used to determine the association between pre-donation zinc protoporphyrin levels and post-transfusion recovery along with the effect of treatment on zinc protoporphyrin levels.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Median (Inter-Quartile Range); unit: μMol/mol heme
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
μMol/mol heme | 54 [47 to 65] | 102 [80 to 136]

3. Secondary Outcome: Serum Ferritin
Description: Measured in a clinical laboratory. Will be used to determine the association between pre-donation ferritin levels and post-transfusion recovery along with the effect of treatment on ferritin levels.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
ug/L | 25.1 [20.4 to 39.6] | 8.4 [6.3 to 10.5]

4. Secondary Outcome: Hemoglobin
Description: Measured in a clinical laboratory. Will be used to determine the association between pre-donation hemoglobin levels and post-transfusion recovery along with the effect of treatment on hemoglobin levels.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
g/dL | 13.9 [12.9 to 14.4] | 11.2 [10.2 to 12.7]

5. Secondary Outcome: Reticulocyte Hemoglobin
Description: Measured in a clinical laboratory. Will be used to determine the association between pre-donation reticulocyte hemoglobin levels and post-transfusion recovery along with the effect of treatment on reticulocyte hemoglobin levels.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
g/dL | 33.2 [32.3 to 34.5] | 29.0 [25.8 to 31.6]

6. Secondary Outcome: Soluble Transferrin Receptor
Description: Measured in a clinical laboratory. Will be used to determine the association between pre-donation soluble transferrin receptor levels and post-transfusion recovery along with the effect of treatment on soluble transferrin receptor levels.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
mg/L | 3.6 [3.2 to 4.5] | 7.0 [5.2 to 9.6]

7. Secondary Outcome: Hepcidin
Description: Measured as a research use only test in a research laboratory using an ELISA from Intrinsic LifeSciences. Will be used to determine the association between pre-donation hepcidin levels and post-transfusion recovery along with the effect of treatment on hepcidin levels.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
ng/mL | 20.3 [16.2 to 31.6] | 15.5 [13.7 to 18.8]

8. Secondary Outcome: Transferrin Saturation
Description: Measured in a clinical laboratory. Will be used to determine the association between pre-donation transferrin saturation levels and post-transfusion recovery along with the effect of treatment on transferrin saturation levels.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
percent | 18.8 [15.1 to 28.5] | 9.1 [7.0 to 13.7]

9. Secondary Outcome: SF-36 Physical Functioning Score
Description: Evaluating subjects' health status using Short Form (SF)-36 question survey. Scores range from 0-100% with higher scores indicating better health.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
percent | 94.83 [91.62 to 98.04] | 94.87 [91.74 to 98.00]

10. Secondary Outcome: SF-36 Role Functioning/Physical Score
Description: as for outcome 9
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
percent | 91.29 [83.87 to 98.7] | 90.36 [83.15 to 97.57]

11. Secondary Outcome: SF-36 Role Functioning/Emotional Score
Description: as for outcome 9
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
percent | 85.58 [75.3 to 95.86] | 81.9 [71.9 to 91.9]

12. Secondary Outcome: SF-36 Energy/Fatigue Score
Description: as for outcome 9
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
percent | 65.94 [59.5 to 72.38] | 61.30 [55.0 to 67.59]

13. Secondary Outcome: SF-36 Emotional Well-being Score
Description: as for outcome 9
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
percent | 79.2 [73.6 to 84.8] | 76.7 [71.2 to 82.2]

14. Secondary Outcome: SF-36 Social Functioning Score
Description: as for outcome 9
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (Inter-Quartile Range); unit: percent
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
percent | 90.7 [84.5 to 96.9] | 87.97 [81.9 to 94.0]

15. Secondary Outcome: SF-36 Pain Score
Description: as for outcome 9
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
percent | 86.9 [81.3 to 92.5] | 88.2 [82.8 to 93.7]

16. Secondary Outcome: SF-36 General Health Score
Description: as for outcome 9
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
percent | 80.3 [74.3 to 86.3] | 73.0 [67.0 to 78.9]

17. Secondary Outcome: SF-36 Health Change Score
Description: as for outcome 9
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
percent | 61.3 [55.4 to 67.2] | 54.6 [48.8 to 60.4]

18. Secondary Outcome: Beck Depression Inventory (BDI) II Score
Description: Evaluating subjects' depression using the Beck Depression Inventory-II survey. Scores range from 0-63 with higher scores indicating more severe depression.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
score on a scale | 4.4 [2.0 to 6.9] | 4.8 [2.4 to 7.2]

19. Secondary Outcome: Beck Anxiety Inventory (BAI) Score
Description: Evaluating subjects' anxiety using the Beck Anxiety Inventory survey. Scores range from 0-63 with higher scores indicating more severe anxiety.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
score on a scale | 3.7 [1.1 to 6.3] | 6.4 [3.8 to 8.9]

20. Secondary Outcome: Global Fatigue Index (GFI) Score
Description: Evaluating subjects' fatigue using the Multidimensional Assessment of Fatigue (MAF) survey. Scores range from 1-50 with higher scores indicating more severe fatigue.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
score on a scale | 11.0 [7.4 to 14.5] | 13.9 [10.4 to 17.4]

21. Secondary Outcome: Restless Legs Syndrome Rating Scale Score
Description: Evaluating subjects' symptoms of restless leg syndrome using the Restless Legs Syndrome Rating Scale survey. Scores range from 0-40 with higher scores indicating more severe symptoms.
Time Frame: End of participation (e.g., ~6 months)
Population: See participant flow for secondary outcomes for subject number explanation.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Iron Repletion | Placebo
Number analyzed (Participants) | 33 | 35
score on a scale | .48 [-0.44 to 1.39] | 1.06 [.16 to 2.0]

ADVERSE EVENTS:
Time Frame: Approximately 6 months of study participation, from first blood donation until final blood draw.
Arm/Group | Iron Repletion | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/40
Other Adverse Events (participants affected / at risk) | 1/39 | 3/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Repletion (N=39) | Placebo (N=40)
cardiac stent (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Repletion (N=39) | Placebo (N=40)
paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT02889133/Prot_SAP_000.pdf